CLINICAL TRIAL: NCT06109818
Title: A Randomized, Double-blind, Placebo-controlled Phase II Clinical Study Evaluating the Efficacy, Safety, Pharmacokinetics, and Pharmacodynamics of ICP-488 in Patients with Moderate to Severe Plaque Psoriasis
Brief Title: Efficacy, Safety, Pharmacokinetics and Pharmacodynamics of ICP-488 in Patients with Moderate to Severe Plaque Psoriasis
Status: Completed | Phase: Phase 2 | Type: Interventional
Sponsor: Beijing InnoCare Pharma Tech Co., Ltd. (Industry)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: Quadruple | Purpose: Treatment
Other Study IDs: ICP-CL-01002
Record Dates: First submitted 2023-10-26; First posted 2023-10-31 (Actual); Last update posted 2025-02-28 (Actual); Status verified 2025-02

CONDITIONS: Moderate to Severe Plaque Psoriasis

STUDY DESIGN:
Who Masked: Participant, Care Provider, Investigator, Outcomes Assessor
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No | US Export: No

ARMS (3):
- ICP-488 low dose (Experimental)
  Interventions: Drug: ICP-488 Tablets; Drug: ICP-488 Placebo
- ICP-488 high dose (Experimental)
  Interventions: Drug: ICP-488 Tablets
- Placebo (Placebo Comparator)
  Interventions: Drug: ICP-488 Placebo

INTERVENTIONS:
Drug: ICP-488 Tablets — ICP-488 will be administered as tablet
  Arms: ICP-488 high dose; ICP-488 low dose
Drug: ICP-488 Placebo — ICP-488 Placebo will be administered as tablet
  Arms: ICP-488 low dose; Placebo

SUMMARY:
This is a multicenter, randomized, double-blind, placebo-controlled Phase II clinical study to evaluate ICP-488.Efficacy, safety, PK, and PD characteristics in Chinese adults with moderate to severe plaque psoriasis.

ELIGIBILITY:
Inclusion Criteria:

1. Subjects voluntarily participate in this study and have signed informed consent.
2. Male or female subjects between the ages of 18 and 70 (including the threshold) at the time of signing the ICF.
3. History of plaque psoriasis ≥6 months at baseline.
4. Subjects need to receive systemic therapy and/or phototherapy.
5. The following three criteria were met: a) psoriasis Area and Severity index (PASI) score ≥12; b) Psoriasis affected body surface area (BSA) ≥10%; c) Static physician overall assessment (sPGA) ≥3 scores

Exclusion Criteria:

1. The diagnosis was non-plaque psoriasis.
2. Presence of infection or immune-related disease.
3. Subjects with a history of TB or at risk for TB.
4. Received related treatment within the time window specified in the protocol.
5. An interval of less than 5 half-lives or 28 days (if any available halflife data) from the last dose of a strong CYP1A2 inhibitor or inducer, or a plan to use concurrently medications, dietary supplements or food with strong CYP1A2 inhibitory or inductive effect during study participation.
6. The investigator has determined that there are clinically significant test results and that participation in this trial would pose an unacceptable risk to patients; Or the laboratory values of the subjects in the screening period meet the criteria specified in the protocol.
7. Pregnant or lactating women, or women who plan to become pregnant during study participation.
8. A history of severe drug allergies.
9. Any other conditions in which the investigator considers it unsuitable for the subject to participate in this study.

Ages: 18 Years to 70 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 129 (Actual)
Dates: Start 2024-01-04 (Actual); Primary Completion 2024-08-05 (Actual); Study Completion 2024-09-18 (Actual)

PRIMARY OUTCOMES:
Percentage of subjects who achieved a PASI 75 response (a reduction of minimum 75% from baseline in PASI score) at Week 12. | Baseline up to Week 12
  Proportion of subjects who achieved PASI 75 (PASI score improvement of at least 75% from baseline) at week 12.

CONTACTS AND LOCATIONS:
Locations (31):
- China (31):
  - Beijing Friendship Hospital, Capital Medical University, Beijing, Beijing Municipality
  - China-Japan Friendship Hospital, Beijing, Beijing Municipality
  - The First Affiliated Hospital of Chongqing Medical University, Chongqing, Chongqing Municipality
  - The First Affiliated Hospital of Fujian Medical University, Fuzhou, Fujian
  - Dermatology Hospital of Southern Medical University, Guangzhou, Guangdong
  - Guangdong Hospital of Traditional Chinese Medicine, Guangzhou, Guangdong
  - Affiliated Hospital of Guizhou Medical University, Guiyang, Guizhou
  - The Affiliated Hospital of Chengde Medical College, Chengde, Hebei
  - The first hospital of hebei medical university, Shijiazhuang, Hebei
  - The Second Affiliated Hospital of Hebei Medical University, Shijiazhuang, Hebei
  - Nanyang city first People's Hospital, Nanyang, Henan
  - Henan Provincial People's Hospital, Zhengzhou, Henan
  - Shiyan City People's Hospital, Shiyan, Hubei
  - Wuhan University People's Hospital, Wuhan, Hubei
  - Wuhan No.1 hospital, Wuhan, Hubei
  - Xiangya hospital central south university, Changsha, Hunan
  - Affiliated Hospital of Inner Mongolia Medical University, Hohhot, Inner Mongolia
  - Changzhou First People's Hospital, Changzhou, Jiangsu
  - Lianyungang First People's Hospital, Lianyungang, Jiangsu
  - Hospital for Skin Diseases, Institute of Dermatology, Chinese Academy of medical Sciences, Peking Union Medical College, Nanjing, Jiangsu
  - First Hospital of Jilin University, Changchun, Jilin
  - Mei he kou central hospital, Meihekou, Jilin
  - Central Hospital affiliated to shandong first medical unversity, Jinan, Shandong
  - Shanghai Dermatology Hospital, Shanghai, Shanghai Municipality
  - Huashan Hospital Affiliated to Fudan University, Shanghai, Shanghai Municipality
  - Chengdu Second People's Hospital, Chengdu, Sichuan
  - The First Affiliated Hospital of Kunming Medical University, Kunming, Yunnan
  - Hangzhou First People's Hospital, Hangzhou, Zhejiang
  - Zhejiang Provincial People's Hospital, Hangzhou, Zhejiang
  - The First Hospital of Jiaxing, Jiaxing, Zhejiang
  - The First Affiliated Hospital of Wenzhou Medical University, Wenzhou, Zhejiang

IPD SHARING:
Plan to Share IPD: No